CLINICAL TRIAL: NCT02251548
Title: A Phase II Study of Ibrutinib in Combination With Fludarabine, Cyclophosphamide, and Rituximab (iFCR) in Previously Untreated, Younger Patients With Chronic Lymphocytic Leukemia
Brief Title: A Phase II Study of Ibrutinib Plus FCR in Previously Untreated, Younger Patients With Chronic Lymphocytic Leukemia
Acronym: iFCR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pharmacyclics LLC. (Industry); The Leukemia and Lymphoma Society (Other); Blood Cancer Research Partnership (Other)
Responsible Party: Principal Investigator, Matthew S. Davids, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-296
Record Dates: First submitted 2014-09-23; First posted 2014-09-29 (Estimated); Results first posted 2020-05-15 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: Chronic lymphocytic leukemia; Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — ibrutinib; fludarabine; fludarabine phosphate; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibrutinib (Experimental): - Ibrutinib-
  * Oral, daily during each cycle
  * fludarabine-administered at standard dosing for up to 6 cycles
  * cyclophosphamide-administered at standard dosing for up to 6 cycles
  * rituximab-administered at standard dosing for up to 6 cycles
  Interventions: Drug: Ibrutinib; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Oral BTK inhibitor
  Other Names: Imbruvica™
Drug: Fludarabine — IV purine analogue chemotherapy agent
  Other Names: Fludara
Drug: Cyclophosphamide — IV alkylator chemotherapy agent
  Other Names: Cytoxan®; Neosar®
Drug: Rituximab — IV anti-CD20 monoclonal antibody
  Other Names: Rituxan®

SUMMARY:
This research study is evaluating a new drug called ibrutinib in combination with the standard drugs fludarabine, cyclophosphamide, and rituximab (FCR) as a possible treatment for Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
Ibrutinib is a type of drug called a kinase inhibitor. It is believed to block a protein called Bruton's tyrosine kinase (BTK) that helps CLL cells live and grow. By blocking this, it is possible that the study drug will kill cancer cells or stop them from growing. Ibrutinib has been FDA approved for the treatment of CLL patients who have received at least one prior treatment; however, the FDA has not yet approved ibrutinib as the first treatment for previously untreated CLL. Therefore, ibrutinib is still considered to be study drug, which means it is still being studied.

Fludarabine, cyclophosphamide, and rituximab (FCR) are intravenous chemotherapy and antibody drugs that together are a standard chemotherapy regimen used for younger patients with CLL. Although FCR is highly effective, it does not typically lead to cure.

In this research study, the investigators are combining a new treatment for CLL, ibrutinib, with a standard chemotherapy regimen for CLL, FCR, to determine whether this combination (iFCR) is safe and effective for patients with previously untreated CLL.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of chronic lymphocytic leukemia or small lymphocytic lymphoma. as per IW-CLL 2008 criteria. Patients must also require therapy for that diagnosis, based on meeting at least one of the following criteria:
* evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia (hemoglobin <11.0 g/L) and/or thrombocytopenia (platelets <100 x 10^9/L)
* massive (≥ 6 cm below the left costal margin), progressive, or symptomatic splenomegaly
* massive nodes (at least 10 cm longest diameter), progressive, or symptomatic lymphadenopathy
* progressive lymphocytosis with an increase of more than 50% over a 2-month period or LDT of <6 months. Lymphocyte doubling time may be obtained by linear regression extrapolation of absolute lymphocyte counts obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In subjects with initial blood lymphocyte counts of <30 x 10^9/L, LDT should not be used as a single parameter to define indication for treatment. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL (eg, infections) should be excluded
* autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy
* documented constitutional symptoms, defined as 1 or more of the following disease-related symptoms or signs:

  * unintentional weight loss >10% within 6 months prior to screening
  * significant fatigue (inability to work or perform usual activities)
  * fevers >100.5° F or 38.0° C for 2 or more weeks prior to screening without evidence of infection
  * night sweats for more than 1 month prior to screening without evidence of infection

    * No prior CLL-directed therapy that was instituted due to patient previously meeting IW-CLL 2008 criteria for treatment
    * Age greater than or equal to 18 years and less than or equal to 65. Because CLL is extremely rare in persons <18 years of age, children are excluded from this study. Because iFCR is an aggressive therapy that is likely to be less well-tolerated even in fit elderly subjects, persons > 65 years of age are excluded
    * ECOG performance status ≤ 1
    * Adequate hematologic function independent of growth factor support for at least 7 days prior to screening and randomization, with the exception of pegylated G-CSF (pegfilgrastim) and darbepoetin which cannot be administered within 14 days of screening.
* Patients must meet the following hematologic criteria at screening:

  * Absolute neutrophil count ≥ 750 cells/mm3 (0.75 x 109/L).
  * Platelet count ≥ 50,000 cells/mm3 (50 x 109/L).
  * Hemoglobin ≥ 8 g/L - Adequate hepatic and renal function defined as:
* Serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN)

  * Bilirubin ≤ 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
  * Adequate renal function defined by serum creatinine >1.5 x ULN
  * PT/INR <1.5 x ULN and PTT (aPTT) <1.5 x ULN.
  * The effects of ibrutinib on the developing human fetus are unknown. For this reason and because similar agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Concurrent Conditions:
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc., or chronic administration of >20 mg/day of prednisone) within 28 days of the first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Recent infection requiring systemic treatment that was completed ≤ 14 days before the first dose of study drug.
* Known bleeding disorders (eg, von Willebrand's disease) or hemophilia.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV). Patients who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Any uncontrolled active systemic infection.
* Major surgery within 4 weeks of first dose of study drug.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Lactating or pregnant.
* Patients receiving any other study agents
* Patients with known CNS involvement
* Baseline QTcF >480 ms. NOTE: This criterion does not apply to patients with a left bundle branch block.
* Patients who require warfarin or other vitamin K antagonists for anticoagulation (other anticoagulants are allowed after consultation with the Principal Investigator).
* Concurrent administration of medications or foods that are strong inhibitors or inducers of CYP3A
* Patients with ongoing use of prophylactic antibiotics are eligible as long as there is no evidence of active infection and the antibiotic is not included on the list of prohibited medications
* Significant co-morbid condition or disease which in the judgment of the Principal Investigator would place the patient at undue risk or interfere with the study
* Unable to receive prophylactic treatment for pneumocystis
* Patients with del(17p) confirmed by FISH in ≥20% of cells or on stimulated karyotype3.2.24 Patients with del(17p) confirmed by FISH in ≥20% of cells or on stimulated karyotype
* Patients with unmutated IGHV who also have a complex karyotype on a stimulated karyotype

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2027-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davids, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (9):
- United States (9):
  - University of Miami Sylvester Comprehensive Cancer Center, Coral Gables, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Deerfield Beach, Florida
  - Unversity of Miami Sylvester Comprehensve Cancer Center, Miami, Florida
  - University of Kansas Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahn IE, Brander DM, Ren Y, Zhou Y, Tyekucheva S, Walker HA, Black R, Montegaard J, Alencar A, Shune L, Omaira M, Jacobson CA, Armand P, Ng SY, Crombie J, Fisher DC, LaCasce AS, Arnason J, Hochberg EP, Takvorian RW, Abramson JS, Brown JR, Davids MS. Five-year follow-up of a phase 2 study of ibrutinib plus fludarabine, cyclophosphamide, and rituximab as initial therapy in CLL. Blood Adv. 2024 Feb 27;8(4):832-841. doi: 10.1182/bloodadvances.2023011574. PMID 38163317
- [Derived] Davids MS, Brander DM, Kim HT, Tyekucheva S, Bsat J, Savell A, Hellman JM, Bazemore J, Francoeur K, Alencar A, Shune L, Omaira M, Jacobson CA, Armand P, Ng S, Crombie J, LaCasce AS, Arnason J, Hochberg EP, Takvorian RW, Abramson JS, Fisher DC, Brown JR; Blood Cancer Research Partnership of the Leukemia & Lymphoma Society. Ibrutinib plus fludarabine, cyclophosphamide, and rituximab as initial treatment for younger patients with chronic lymphocytic leukaemia: a single-arm, multicentre, phase 2 trial. Lancet Haematol. 2019 Aug;6(8):e419-e428. doi: 10.1016/S2352-3026(19)30104-8. Epub 2019 Jun 14. PMID 31208944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to enrollment on 10/3/2014 and closed to enrollment on 4/24/2018. 58 participants were enrolled at Dana-Farber, 9 at Massachusetts General Hospital, 3 at Beth Israel Deaconess Medical Center, 9 at Duke University, 1 at University of Kansas, 3 at West Michigan Cancer Center, and 2 at University of Miami for a total of 85 enrolled.
Groups:
- FCR +420mg Ibrutinib Daily: Patients received oral agent ibrutinib daily on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day ibrutinib run in, then will continue daily dosing.Fludarabine, cyclophosphamide, rituximab (FCR) will be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients will receive ibrutinib monotherapy indefinitely unless they are found to be minimal residual disease(MRD) negative in the bone marrow at the 24 months of ibrutinib maintenance timepoint, at which point they will discontinue ibrutinib to undergo active disease monitoring. If during active monitoring they develop MRD positivity in the blood, they may resume ibrutinib monotherapy. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities
Period: Overall Study
Arm/Group | FCR +420mg Ibrutinib Daily
Started | 85
Completed | 0
Not Completed | 85

BASELINE CHARACTERISTICS:
Population: Age greater than or equal to 18 years and less than or equal to 65 with no prior CLL directed therapy that was instituted due to patient previously meeting IWCLL 2008 criteria for treatment
Groups:
- FCR+ 420 mg Ibrutinib daily: Patients received oral agent ibrutinib daily on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day ibrutinib run in, then will continue daily dosing.Fludarabine, cyclophosphamide, rituximab (FCR) will be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients will receive ibrutinib monotherapy indefinitely unless they are found to be minimal residual disease(MRD) negative in the bone marrow at the 24 months of ibrutinib maintenance timepoint, at which point they will discontinue ibrutinib to undergo active disease monitoring. If during active monitoring they develop MRD positivity in the blood, they may resume ibrutinib monotherapy. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants] — Participants were eligible if their age was greater than or equal to 18 years and less than or equal to 65
  Participants
    <=18 years | 0
    Between 18 and 65 years | 85
    >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 55 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 82
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants] — Enrolled in the United States of America
  Participants
    United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Part I: Participants Who Achieve a Minimal Residual Disease (MRD) Negative Complete Response (CR) in the Bone Marrow at 2 Months Post FCR
Description: To assess the number of participants who achieve an MRD negative complete response at the 2 months post last dose of FCR timepoint by 2008 IW-CLL criteria ( Hallek et. al). Participants will have a bone marrow biopsy procedure 2 months after completing combination therapy (Ibrutinib+ FCR) in tandem with a chest, neck, abdomen and pelvic PET CT scan. A central read of the PET CT scan will confirm a radiographic complete response, and the bone marrow pathology and morphology assessments will confirm morphological CR in the bone marrow, while MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4.
Time Frame: 2 months after completing combination therapy
Population: No prior CLL-directed therapy that was instituted due to patient previously meeting IWCLL 2008 criteria for treatment- Age greater than or equal to 18 years and less than or equal to 65 and must require therapy by standard IW-CLL 2008 criteria with adequate renal, hepatic, and hematologic function
Measure: Count of Participants; unit: Participants
Groups:
- FCR+ 420mg Ibrutinib Daily: Patients received oral agent ibrutinib daily on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day ibrutinib run in, then will continue daily dosing.Fludarabine, cyclophosphamide, rituximab (FCR) will be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients will receive ibrutinib monotherapy indefinitely unless they are found to be minimal residual disease(MRD) negative in the bone marrow at the 24 months of ibrutinib maintenance timepoint, at which point they will discontinue ibrutinib to undergo active disease monitoring. If during active monitoring they develop MRD positivity in the blood, they may resume ibrutinib monotherapy. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities
Arm/Group | FCR+ 420mg Ibrutinib Daily
Number analyzed (Participants) | 85
Participants | 28

2. Primary Outcome: Part II: Participants Who Achieve a Minimal Residual Disease (MRD) Negative Complete Response (CR) in the Bone Marrow at 2 Years Post Discontinuation of Ibrutinib After Having Achieved MRD Negative CR at the 2 Months Post FCR Timepoint
Description: Participants will have bone marrow biopsies in tandem with a chest, neck, abdomen and pelvic PET CT scan as clinically indicated after discontinuation of treatment. A central read of the PET CT scan will confirm the radiographic response, and the bone marrow pathology and morphology assessments will confirm morphological response in the bone marrow, while MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008).
Time Frame: 2 years post discontinuation of ibrutinib after 24 months of ibrutinib maintenance
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Overall Response Rate
Description: The objective response rate (ORR) was defined as the proportion of participants achieving CR+CRi+PR, Complete Response with incomplete count recovery (CRi) or partial response (PR) based on 2008 IW-CLL criteria criteria (Hallek et al., 2008).
Time Frame: Response evaluated at 2 months post iFCR. Treatment up to 6 cycles (28 days each).
Measure: Number; unit: proportion of participants
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 85
proportion of participants | 0.96

4. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR defined as the proportion of participants achieving complete response. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008).
Time Frame: Response evaluated at 2 months post iFCR. Treatment up to 6 cycles (28 days each).
Measure: Number; unit: proportion of participants
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 85
proportion of participants | 0.24

5. Secondary Outcome: Partial Response Rate (PRR)
Description: PRR defined as the proportion of participants achieving partial response. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008).
Time Frame: Response evaluated at 2 months post iFCR. Treatment up to 6 cycles (28 days each).
Measure: Number; unit: proportion of participant
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 85
proportion of participant | 0.61

6. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last dsease assessment.
Time Frame: Disease will be evaluated through imaging cycle 3-6 day 1, and In long-term follow-up, after removal or until participant withdrawal, death, or removal from study. Median follow-up is: 63.24 months (range: 6.83-95.8).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 85
months | NA [NA to NA] — insufficient number of participants with events

7. Secondary Outcome: Median Overall Survival (OS)
Description: Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Median follow-up is: 63.24 months (range: 6.83-95.8).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 85
months | NA [NA to NA] — insufficient number of participants with events

8. Secondary Outcome: Rate of MRD Negative CR After 3 Cycles of iFCR
Description: To determine the rate of minimal residual disease negative complete response (MRD negative CR) in the bone marrow after 3 cycles of ibrutinib + FCR. Participants will have a bone marrow biopsy procedure after completing 3 cycles in tandem with a chest, neck, abdomen and pelvic PET CT scan. A central read of the PET CT scan will confirm a radiographic complete response, and the bone marrow pathology and morphology assessments will confirm morphological CR in the bone marrow, while MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)
Time Frame: After 3 cycles of iFCR for each patient completing 3 cycles
Measure: Count of Participants; unit: Participants
Groups:
- FCR +420mg Ibrutinib Daily: Patients received oral agent ipilimumab daily on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day ipilimumab run in, then will continue daily dosing.Fludarabine, cyclophosphamide, rituximab (FCR) will be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients will receive ibrutinib monotherapy indefinitely unless they are found to be minimal residual disease(MRD) negative in the bone marrow at the 24 months of ibrutinib maintenance timepoint, at which point they will discontinue ibrutinib to undergo active disease monitoring. If during active monitoring they develop MRD positivity in the blood, they may resume ibrutinib monotherapy. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities
Arm/Group | FCR +420mg Ibrutinib Daily
Number analyzed (Participants) | 85
Participants | 9

9. Secondary Outcome: 1-year Combined Response With MRD From Bone Marrow
Description: Combined response with MRD from bone marrow reported as the MRD-negative CR. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)
Time Frame: at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 85
Participants | 2

10. Secondary Outcome: Number of Participants Who Convert From Bone Marrow MRD Negative PR to Bone Marrow MRD Negative CR After 1 Year of Ibrutinib Maintenance
Description: To determine the rate of minimal residual disease negative complete response (MRD negative CR) in the bone marrow at 12 months from start of therapy, participants will have a bone marrow biopsy procedure at the 1 year timepoint after completing combination therapy (ibrutinib + FCR) in tandem with a chest, neck, abdomen and pelvic PET CT scan. A central read of the PET CT scan will confirm a radiographic complete response, and the bone marrow pathology and morphology assessments will confirm morphological CR in the bone marrow, while MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)
Time Frame: 12 months ( 1year) after starting therapy
Measure: Count of Participants; unit: Participants
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 40
Participants | 2

11. Secondary Outcome: Number of Participants Who Convert From Bone Marrow MRD Negative PR to Bone Marrow MRD Negative CR After 2 Years on Treatment
Description: MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)- Bone marrow biopsies will be performed at baseline, after cycle 3, 2 months post FCR, at 1 year and 2 years of ibrutinib maintenance, and as clinically indicated thereafter- Participants will have a bone marrow biopsy procedure 24 months after completing combination therapy (Ibrutinib+ FCR) in tandem with a chest, neck, abdomen and pelvic PET CT scan. A central read of the PET CT scan will confirm a radiographic complete response, and the bone marrow pathology and morphology assessments will confirm morphological CR in the bone marrow, while MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4.
Time Frame: 2 years (24 months) from start of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 40
Participants | 9

12. Secondary Outcome: Median Time to Bone Marrow MRD Negativity
Description: MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)-
Time Frame: Bone marrow biopsies will be performed at baseline, after cycle 3, 2 months post FCR, at 1 year and 2 years of ibrutinib maintenance, and as clinically indicated thereafter
Measure: Median (Full Range); unit: months
Arm/Group | FCR+ 420 mg Ibrutinib daily
Number analyzed (Participants) | 71
months | 3 [2.79 to 23.69]

13. Secondary Outcome: Participants Who Convert From Bone Marrow MRD Negativity to MRD Positivity in Participants Who Discontinue Ibrutinib
Description: .MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4. Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)
Time Frame: Response evaluated at 2 months post iFCR. Treatment up to 6 cycles (28 days each).
Measure: Count of Participants; unit: Participants
Groups:
- FCR+Ibrutinib 420mg Daily: Patients received oral agent ipilimumab daily on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day ipilimumab run in, then will continue daily dosing. Fludarabine, cyclophosphamide, rituximab (FCR) will be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients will receive ibrutinib monotherapy indefinitely unless they are found to be minimal residual disease(MRD) negative in the bone marrow at the 24 months of ibrutinib maintenance timepoint, at which point they will discontinue ibrutinib to undergo active disease monitoring. If during active monitoring they develop MRD positivity in the blood, they may resume ibrutinib monotherapy. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities
Arm/Group | FCR+Ibrutinib 420mg Daily
Number analyzed (Participants) | 33
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events are assessed from the time the participants sign informed consent, and then are assessed by the study team at minimum every week during cycle 1, and day 1 of every cycle thereafter during combination, then every three cycles thereafter while in maintenance for the duration of their time on active treatment through study completion, an average of 3 years. Intra-cycle communication occurs throughout the treatment phase of the trial by electronic medical record secure email.
Description: Maximum grade toxicity by type-Serious AEs were defined as per DFCI criteria: Any grade 2, 3, or 4 unexpected and treatment related event, and all and 5 events regardless of attribution to study treatment , and includes events deemed medically important by overall PI. Other AEs were defined as events with the attribution of at least possibly related to the study treatment that did not meet the SAE criteria. CTCAE 4.0 was used in investigator assessment and lab value review.
Arm/Group | FCR+Ibrutinib 420mg Daily
All-Cause Mortality (participants affected / at risk) | 1/85
Serious Adverse Events (participants affected / at risk) | 24/85
Other Adverse Events (participants affected / at risk) | 85/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR+Ibrutinib 420mg Daily (N=85)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Lipase Increased (Investigations) | 1 (1)
Alanine Amintransferase Increased (Investigations) | 3 (3)
Appendicitis (Infections and infestations) | 1 (1)
Anaplasmosis (Infections and infestations) | 1 (1)
Pneumatosis (Gastrointestinal disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-Cardiac Chest Pain (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Pneumocystis Jivrocii Pneumonia (Infections and infestations) | 3 (3)
Secondary Malignancy- Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sudden Death (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Respiratory Syncytial Virus (Infections and infestations) | 1 (1)
Appendiceal Mucocele (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) — MRSA; Septic Shock
Hemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FCR+Ibrutinib 420mg Daily (N=85)
Rash acneiform (Skin and subcutaneous tissue disorders) | 26
Aspartate aminotransferase increased (Investigations) | 25
Hyponatremia (Metabolism and nutrition disorders) | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23
Headache (Nervous system disorders) | 21
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 21
Lymphocyte count increased (Investigations) | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 20
Leukocytosis (Blood and lymphatic system disorders) | 18
Upper respiratory infection (Infections and infestations) | 18
Vomiting (Gastrointestinal disorders) | 18
Alanine aminotransferase increased (Investigations) | 17
Fever (General disorders and administration site conditions) | 17
Hyperkalemia (Metabolism and nutrition disorders) | 17
Insomnia (Psychiatric disorders) | 17
Blood bilirubin increased (Investigations) | 16
Gastroesophageal reflux disease (Gastrointestinal disorders) | 15
Hypokalemia (Metabolism and nutrition disorders) | 15
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 13
Dry skin (Skin and subcutaneous tissue disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 13
Anxiety (Psychiatric disorders) | 12
Dizziness (Nervous system disorders) | 12
Edema limbs (General disorders and administration site conditions) | 12
Palpitations (Cardiac disorders) | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11
Alkaline phosphatase increased (Investigations) | 10
Dyspepsia (Gastrointestinal disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 10
Creatinine increased (Investigations) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Lung infection (Infections and infestations) | 9
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 9
Pain (General disorders and administration site conditions) | 9
Abdominal pain (Gastrointestinal disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Chills (General disorders and administration site conditions) | 7
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 7
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Hot flashes (Vascular disorders) | 6
Hypertension (Vascular disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 6
Sinusitis (Infections and infestations) | 6
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Atrial fibrillation (Cardiac disorders) | 5
Depression (Psychiatric disorders) | 5
Dry mouth (Gastrointestinal disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Hypernatremia (Metabolism and nutrition disorders) | 5
Infusion related reaction (General disorders and administration site conditions) | 5
Investigations - Other, specify (Investigations) | 5
Localized edema (General disorders and administration site conditions) | 5
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT02251548/Prot_SAP_000.pdf